CLINICAL TRIAL: NCT00769613
Title: Emergency Access to C.V. pp65 / IE-1 Specific Cytotoxic T Lymphocytes for Recipients of Allogeneic Stem Cell Transplants With Persistant or Therapy Refractory Infections
Brief Title: Emergency Use of Donor Lymphocytes in Treating Patients Who Have Undergone Donor Stem Cell Transplant and Have Cytomegalovirus Infections
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000615167; PSCI-PSHCI-08-051
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2010-08

CONDITIONS: Cancer
Keywords: stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL1 negative; blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; juvenile myelomonocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; childhood myelodysplastic syndromes; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; myelodysplastic/myeloproliferative neoplasm, unclassifiable; high risk metastatic gestational trophoblastic tumor; previously treated childhood rhabdomyosarcoma; previously treated myelodysplastic syndromes; recurrent Wilms tumor and other childhood kidney tumors; recurrent childhood rhabdomyosarcoma; recurrent neuroblastoma; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent malignant testicular germ cell tumor; secondary myelodysplastic syndromes; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; refractory multiple myeloma; cytomegalovirus infection
MeSH Terms: conditions — Neoplasms; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Recurrence; Mycosis Fungoides; Sezary Syndrome; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Leukemia, Myeloid, Acute; Leukemia, Hairy Cell; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Myeloproliferative Disorders; Wilms Tumor; Neuroblastoma; Carcinoma, Ovarian Epithelial; Testicular Neoplasms; Multiple Myeloma; Breast Neoplasms; Cytomegalovirus Infections | interventions — Polymerase Chain Reaction; Flow Cytometry

INTERVENTIONS:
Biological: cytomegalovirus IE-1-specific cytotoxic T lymphocytes
Biological: cytomegalovirus pp65-specific cytotoxic T lymphocytes
Biological: therapeutic allogeneic lymphocytes
Genetic: polymerase chain reaction
Other: flow cytometry
Other: immunological diagnostic method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: White blood cells that have been treated in the laboratory may kill cells that are infected with cytomegalovirus.

PURPOSE: This phase I trial is studying how well cytotoxic T cells work in treating patients who have undergone donor stem cell transplant and have cytomegalovirus infections.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To provide access to cytomegalovirus (CMV) pp65- and IE-1-specific cytotoxic T lymphocytes (CTL) in patients with persistent CMV infections after allogeneic stem cell transplantation.

Secondary

* To characterize CMV pp65- and IE-1-specific immune responses in terms of cytotoxicity and cytokine production pre-infusion and then periodically thereafter.
* To characterize the levels of CMV DNA in recipients of CMV pp65- and IE-1-specific CTL and observe whether the CTL infusion has any impact on level of virus.
* To determine the feasibility of CMV CTL culture from CMV-seronegative donors who have received a CMV vaccine.

OUTLINE: This is a multicenter study.

Patients receive allogeneic cytomegalovirus (CMV) pp65- and IE-1-specific cytotoxic T-cell lymphocytes infusion over 5 minutes on day 1. Patients may receive up to 2 more doses at least 2 weeks after previous dose.

Blood samples are collected and analyzed by quantitative CMV PCR, chromium-release assays for CMV pp65- and IE-1-specific cytotoxicity, and immunophenotype for CD3, CD4, CD8, CD56, CD19, and CD45RA/RO. Intracellular cytofluorometry is used to assess IL-2, IL-4, IL-10, and IFN-γ production by CD4 and CD8 CMV-specific effector cells.

After completion of study therapy, patients are followed periodically for up to 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Recipient of an allogeneic stem cell transplantation
* Cytomegalovirus (CMV)-seropositive and meeting 1 of the following criteria:

  * Patient has a history of CMV antigenemia for ≥ 2 weeks
  * CMV DNA levels ≥ 600 copies/mcg of DNA despite antiviral therapy targeting CMV (e.g., ganciclovir or foscarnet)
* No ongoing graft-vs-host disease
* Has donor available for peripheral blood mononuclear cell collection (for cytotoxic T lymphocytes production), meeting either of the following criteria:

  * CMV-seropositive donor (≥ 2 years of age)
  * CMV-seronegative related donor (≥ 18 years of age) who consents to receive the CMV vaccine

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-3 OR Lansky PS 50-100% (for patients < 16 years of age)
* Bilirubin < 2.0 mg/dL
* AST and ALT < 2.5 times normal
* Creatinine clearance ≥ 30 mL/min
* Pulse oximetry ≥ 94% on no more than 40% oxygen by face mask
* Not moribund
* No patients expected to survive ≤ 1 month after the T-cell infusion due to cardiac, pulmonary, renal, hepatic, or neurologic dysfunction

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Must be on ≤ 1 mg/kg/day of prednisone or its equivalent at the time of study CTL infusion

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-08; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Safety
Toxicity

SECONDARY OUTCOMES:
Time to development of cytomegalovirus (CMV)-specific immune reconstitution
CMV DNA levels
Time during post-infusion follow-up at which the dominant CMV pp65- and IE-1 epitopes for the donor is recognized by the cytotoxic T-cell lymphocytes (CTL)
Feasibility of CMV pp65- and IE-1 CTL culture after CMV vaccination of seronegative donors

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G. Lucas, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States